CLINICAL TRIAL: NCT02484638
Title: A Multicenter, Open-label, Multiple-dose, Dose Escalation Study to Investigate the Pharmacokinetics, Efficacy, and Safety of rVIIa-FP (CSL 689) in Subjects With Hemophilia (A or B) and Inhibitors
Brief Title: Study of Recombinant Factor VIIa Fusion Protein (rVIIa-FP, CSL689) for On-demand Treatment of Bleeding Episodes in Patients With Hemophilia A or B With Inhibitors
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Business decision non-safety related.
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSL689_2001; 2012-001309-26 (EudraCT Number)
Record Dates: First submitted 2015-06-25; First posted 2015-06-29 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hemophilia A With Inhibitors; Hemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CSL689 low-dose (Experimental): * Part 1: single injection of low-dose CSL689 for PK evaluation
  * Part 2: up to 2 injections of low-dose CSL689 per bleeding event (bleeding events 1 to 3*)
  * Part 3: up to 3 injections of low-dose CSL689 per bleeding event * Note: All subjects in the low-dose arm will be treated with high-dose CSL689 for bleeding events 4-6 in Part 2
  Interventions: Drug: CSL689
- CSL689 high-dose (Experimental): * Part 1: single injection of high-dose CSL689 for PK evaluation
  * Part 2: up to 2 injections of high-dose CSL689 per bleeding event (bleeding events 4 to 6*)
  * Part 3: up to 3 injections of high-dose CSL689 per bleeding event
    * Note: All subjects in the high-dose arm will be treated with low-dose CSL689 for bleeding events 1-3 in Part 2
  Interventions: Drug: CSL689
- Eptacog alfa low-dose (Active Comparator): Single injection of low-dose Eptacog alfa in Part 1 for PK evaluation
  Interventions: Drug: Eptacog alfa (activated)
- Eptacog alfa high-dose (Active Comparator): Single injection of high-dose Eptacog alfa in Part 1 for PK evaluation
  Interventions: Drug: Eptacog alfa (activated)

INTERVENTIONS:
Drug: CSL689 — Recombinant fusion protein, linking activated coagulation factor VII with albumin. Two dose levels (low dose, high dose) will be studied in Parts 1, 2, and 3.
  Arms: CSL689 high-dose; CSL689 low-dose
Drug: Eptacog alfa (activated) — Recombinant activated coagulation factor VII. Two dose levels (low dose, high dose) will be studied in Part 1.
  Arms: Eptacog alfa high-dose; Eptacog alfa low-dose

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics (PK), efficacy, and safety of rVIIa-FP (CSL689). The study will enroll approximately 54 male subjects, 12 to 65 years of age, with hemophilia types A or B who have developed inhibitors to FVIII or FIX. The study consists of 3 sequential parts (Parts 1, 2, 3): The purpose of Part 1 (PK part) is to evaluate the PK of a single treatment of CSL689 (low dose or high dose) and compare with the PK of a single treatment of Eptacog alfa (low dose or high dose). In Part 1, CSL689 and Eptacog alfa will be given by the doctor at the study center. The purpose of Part 2 (Dose-evaluation part) is to identify which of the 2 tested dose levels of CSL689 shows the best efficacy and safety in stopping acute bleeding events (this dose will be called the "population best dose"). The purpose of the final Part 3 (Repeated-dose part) is to confirm the efficacy and safety of the "population best dose" identified in Part 2. In Parts 2 and 3, subjects will self-administer a specified number of CSL689 infusions at home on-demand (ie, when a bleeding event occurs), will keep an electronic diary, and will visit the center at monthly intervals. This study is expected to last for up to 16 months for the subjects participating in all 3 parts, and up to 9 months for the subjects participating in Part 3 only.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with hemophilia A or B and inhibitors.
* Age ≥ 12 and ≤ 65 years.
* High responding inhibitor with documented historical inhibitor titer > 5 Bethesda Units/mL.

Exclusion Criteria:

* Congenital or acquired coagulation disorders other than hemophilia A or B.
* Ongoing immune tolerance induction therapy or planned during study.
* Known or suspected hypersensitivity to activated recombinant human FVII or to any excipient of CSL689.
* Body mass index > 30 kg/m².
* Major surgery within 28 days before screening or scheduled major and / or orthopedic surgery during the study.
* Advanced atherosclerotic disease (ie, known history of ischemic heart disease, or ischemic stroke).
* Any clinical signs or known history of thromboembolic events, including known deep vein thrombosis.
* Human immunodeficiency virus (HIV)-positive subjects who have low cluster of differentiation 4 (CD4)+ lymphocyte count (200/μL or less) at screening.
* Use of the following within the screening period or planned during study: a) plasma or coagulation factor concentrates other than rescue therapy or therapy during Part 1, b) other platelet inhibitors, c) desmopressin, and d) fibrinolysis inhibitors, except if used as local treatment (eg, for oral bleeds).

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07-23 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC0-t) | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
  Area under plasma factor VIIa activity versus time curve from time 0 to last sample with quantifiable activity (in Part 1 only).
Incremental recovery | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
  Incremental recovery of plasma factor VIIa activity (in Part 1 only)
Elimination half-life | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
  Elimination half-life of plasma factor VIIa activity (in Part 1 only)
Total clearance | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
  Total clearance of plasma factor VIIa activity (in Part 1 only)
Treatment success with first CSL689 injection | Up to 8 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the first injection of CSL689 for each bleeding event in Part 2.
Treatment success with first CSL689 injection at the population best dose | Up to 8 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the first injection of the population best dose of CSL689 in subjects participating only in Part 3, along with its 95% confidence interval
Treatment success with first or second CSL689 injection at the population best dose | Up to 16 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the first or second injection of the population best dose of CSL689 in subjects participating in Part 3 only, along with its 95% confidence interval

SECONDARY OUTCOMES:
Treatment success with first or second CSL689 injection | Up to 16 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the first or second (if required) injection of CSL689 for each bleeding event in Part 2.
Number of bleeding events requiring > 1 CSL689 injection | Up to 8 hours after first CSL689 injection for each bleeding event
  Outcome measure will be analyzed for Part 2 and for Part 3
Number of CSL689 injections per bleeding event | Up to 16 hours (Part 2) or up to 24 hours (Part 3) after first CSL689 injection for each bleeding event
  Outcome measure will be analyzed for Part 2 and for Part 3
Total dose of CSL689 per bleeding event | Up to 16 hours (Part 2) or up to 24 hours (Part 3) after first CSL689 injection for each bleeding event
  Outcome measure will be analyzed for Part 2 and for Part 3
Treatment success with first CSL689 injection at the population best dose | Up to 8 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the first injection of CSL689 for each bleeding event at the population best dose in subjects participating in Part 3
Percentage of first bleeding events successfully treated with first CSL689 injection at population best dose in Part 3 | Up to 8 hours after first CSL689 injection for first bleeding event
Treatment success at population best dose | Up to 24 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the:
  * first or second injection
  * first, second or third injection of the population best dose of CSL689 in Part 3
Treatment success with CSL689 at the dose level that is not the population best dose | Up to 24 hours after first CSL689 injection for each bleeding event
  Percentage of bleeding events successfully treated with the:
  * first injection
  * first or second injection
  * first, second or third injection at the dose level that is not the population best dose of CSL689 in Part 3
Percentage of bleeding events with only "definite" or "abrupt" subject-reported pain relief at the population best dose | Up to 24 hours after CSL689 injection for each bleeding event
Percentage of bleeding events with "good" or "excellent" investigator-reported assessment of treatment response at the population best dose of CSL689 | Up to 9 months
Proportion of recurrences | Up to 9 months
  Recurrence defined as a bleeding in the same joint/anatomical location within 24 hours after an initial "good" or "excellent" response.
Proportion of bleeding events with ultrarapid progression. | Up to 9 months
  "Ultrarapid progression" is defined as overt, uncontrolled hemorrhage and / or progressive increase in pain and / or rapid progression in hematoma size
Proportion of bleeding events requiring post-hemostatic maintenance dosing | Up to 9 months
Number of subjects with treatment-emergent adverse events (TEAEs) | Up to 16 months
  TEAEs are adverse events (AEs) that start on or after the date and time of the first injection of either CSL689 or Eptacog alfa.
  Number of subjects with TEAEs will be presented:
  * Overall
  * Related to CSL689
Percentage of subjects with TEAEs | Up to 16 months
  TEAEs are AEs that start on or after the date and time of the first injection of either CSL689 or Eptacog alfa.
  Percentage of subjects with TEAEs will be presented:
  * Overall
  * Related to CSL689
Number of subjects with an antibody response | Up to 16 months
  Number of subjects with:
  * Inhibitors against FVII
  * Antibodies to CSL689
Percentage of subjects with an antibody response | Up to 16 months
  Percentage of subjects with:
  * Inhibitors against FVII
  * Antibodies to CSL689
AUC(0-inf) | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
  Area under plasma factor VIIa activity versus time curve from time 0 extrapolated to infinity
Maximum observed plasma FVIIa activity (Cmax) | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
Time of occurrence of maximum observed plasma FVIIa activity (Tmax) | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
Volume of distribution at steady state (Vss) | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689
Mean residence time (MRT) | Before injection and at up to 6 time points until 24 hours after injection for Eptacog alfa; before injection and at up to 11 time points until up to 120 hours after injection for CSL689

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — CSL Behring
Locations (10):
- Site Reference # 2680001, Tbilisi, Georgia
- Site Reference # 3800023, Milan, Italy
- Site Reference # 4580001, Kuala Lumpur, Malaysia
- Site Reference # 6430026, Kemerovo, Russia
- Site Reference # 7100001, Johannesburg, South Africa
- Site Reference # 7240007, Madrid, Spain
- Thailand (2):
  - Site Reference # 7640006, Bangkok
  - Site Reference # 7640004, Khon Kaen
- Site Reference # 8040005, Lviv, Ukraine
- Site Reference # 8260008, London, United Kingdom